CLINICAL TRIAL: NCT06142045
Title: Cerebrovascular Responses to Isometric Exercise, and Hypercapnia in Children, Adolescents and Adults
Brief Title: Brain Blood Flow Responses at Rest and During Exercise
Status: Not yet recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Ai McManus, Professor, University of British Columbia
Other Study IDs: H23-02316
Record Dates: First submitted 2023-11-13; First posted 2023-11-21 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Cerebrovascular Regulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Children (7-10 years): All groups of the experiment will be exposed to the same intervention. The intervention the participants are exposed to is the use of the computer controlled gas blender system for manipulation of end-tidal and arterial blood gases. This will be used for the following protocols, to either clamp end-tidal concentrations at resting levels or administer a hypercapnia challenge. The protocol includes assessment of cerebral blood flow responses (measured using ultrasound) to carbon dioxide; including a hypercapnia ramp protocol followed by a transient protocol. Following at least 30 minute wash out, participants will then perform isometric exercise at 30% of their maximal voluntary contraction for 2 minutes. Participants will perform the isometric handgrip exercise under 2 different conditions (hypercapnia (+9 mmHg) and clamped breathing; to maintain baseline end-tidal carbon dioxide and oxygen concentrations) with a 20-minute recovery period between each bout.
  Interventions: Device: RespirACT RA-MR System
- Adolescents (12-16 years): All groups of the experiment will be exposed to the same intervention. The intervention the participants are exposed to is the use of the computer controlled gas blender system for manipulation of end-tidal and arterial blood gases. This will be used for the following protocols, to either clamp end-tidal at resting levels or administer a hypercapnia challenge. The protocol includes assessment of cerebral blood flow responses (measured using ultrasound) to carbon dioxide; including a hypercapnia ramp protocol followed by a transient protocol. Following at least 30 minute wash out, participants will then perform isometric exercise at 30% of their maximal voluntary contraction for 2 minutes. Participants will perform the isometric handgrip exercise under 2 different conditions (hypercapnia (+9 mmHg) and clamped breathing; to maintain baseline end-tidal carbon dioxide and oxygen concentrations) with a 20-minute recovery period between each bout.
  Interventions: Device: RespirACT RA-MR System
- Adults (18-35 years): All groups of the experiment will be exposed to the same intervention. The intervention the participants are exposed to is the use of the computer controlled gas blender system for manipulation of end-tidal and arterial blood gases. This will be used for the following protocols, to either clamp end-tidal at resting levels or administer a hypercapnia challenge. The protocol includes assessment of cerebral blood flow responses (measured using ultrasound) to carbon dioxide; including a hypercapnia ramp protocol followed by a transient protocol. Following at least 30 minute wash out, participants will then perform isometric exercise at 30% of their maximal voluntary contraction for 2 minutes. Participants will perform the isometric handgrip exercise under 2 different conditions (hypercapnia (+9 mmHg) and clamped breathing; to maintain baseline end-tidal carbon dioxide and oxygen concentrations) with a 20-minute recovery period between each bout.
  Interventions: Device: RespirACT RA-MR System

INTERVENTIONS:
Device: RespirACT RA-MR System — RespirAct RA-MR™ is a computer-controlled gas blender to implement precise control of blood gases for a consistent and repeatable stimulus.

SUMMARY:
Tight regulation of brain blood flow is integral for delivery of oxygen and energy for survival. During childhood, the brain has a twofold higher metabolic requirement, thus requires greater blood flow to match this. Despite this knowledge, brain blood flow responses and the mechanisms of regulation during maturation are largely unknown. Thus, we are trying to understand what happens to blood vessel function and the mechanisms of regulation at rest and during handgrip exercise. This will give us valuable information on brain blood vessel responses, which will help future interventions aimed at improving blood vessel function in youth, for future disease prevention. Utilizing the pubertal transition will provide insights into the influence of sex hormones on brain blood flow regulation.

The goal of this cross-sectional observational study is to examine the influence of age and maturation on cerebral blood flow regulation, achieved through exploring the responses to increases in carbon dioxide concentrations, and static handgrip exercise in children (7-10 years), adolescents (12-16 years) and young adults (19-35 years).

The main questions the study aims to answer are:

* Investigate the brain blood flow responses to increases in carbon dioxide concentrations in children, adolescents and adults.
* Investigate brain blood flow responses to handgrip exercise with and without increases in carbon dioxide concentrations in children, adolescents and adults.

During all protocols, participants will have their end-tidal gas concentrations measured and/or altered using prospective end-tidal gas targeting using a computer controlled gas blender system in which we have obtained Health Canada approval for.

DETAILED DESCRIPTION:
The goal of this cross-sectional experimental study to determine the influence age, sex and pubertal status on cerebrovascular responses at rest and during isometric exercise.

The main objective is to investigate the regulatory mechanisms of cerebral blood flow during hypercapnia and isometric exercise, and determine whether any mechanistic differences in regulation are present with advancing age and maturation.

The following questions will be addressed in 20 healthy children (7-10 years), 20 healthy adolescents (12-16 years) and 20 young healthy adults (19-35 years), to compare the influence of age, sex and maturation on these responses, as follows:

1. Investigate the brain blood flow responses to isometric exercise with and without hypercapnia (+9 mmHg carbon dioxide) in children, adolescents and adults.
2. Investigate the brain blood flow responses to hypercapnia (+9 mmHg carbon dioxide) in children, adolescents and adults using a ramp incremental 4 minute protocol compared with a 30 second protocol, to identify which method is the most tolerable in children and adolescents.
3. Determine whether sex, and the sex-dependent influences of age and maturation influence any of the brain blood flow responses to hypercapnia or isometric handgrip exercise.

To control and manipulate breathing gases during the study protocols, the partial pressures of end-tidal carbon dioxide and oxygen will be sampled at the mouth using the Investigational Testing Authorization approved computer controlled gas blender system. To target specific end-tidal carbon dioxide and oxygen levels during the clamped breathing and hypercapnic trials respectively, prospective end-tidal gas targeting will be utilized. The system allows for breath-by-breath regulation of end-tidal gases, independently of ventilation. End-tidal concentrations are prospectively targeted by controlling the inspired concentration of carbon dioxide and oxygen according to the previous expired breath, allowing this to be precisely controlled throughout the duration of the protocol. Gas analysis, and spirometry measures of tidal volume and breathing frequency will be recorded using the computer controlled system. Prospective end-tidal gas targeting is safe, with all inspired gases containing oxygen, with rigorous control procedures and fail-safe mechanisms which do not allow inhaled gases to fall outside of safe thresholds.

ELIGIBILITY:
Inclusion Criteria:

* Are aged between 7-10 years, 12-16 years or 19-35 years
* Male or Female
* Have a normal blood pressure (<160/110 mmHg) and are not taking any anti-hypertensive medications.
* No prior or current history of cardiorespiratory of cerebrovascular diseases.
* Can communicate in English

Exclusion Criteria:

* Inability to perform handgrip exercise
* Are currently taking any medications known to influence vascular function, heart rate or blood pressure
* Have epilepsy
* Are a current smoker
* Have known cardiometabolic abnormalities
* Have congenital cardiac abnormalities (e.g., tetralogy of Fallot)
* Unstable angina (frequent chest pain)
* Atrial Fibrillation
* Myocardial infarction (heart attack) within the previous 3 months
* Transient ischemic attack (TIA) within the previous 6 months
* Heart failure ≥ class 2
* Have a known respiratory disease (e.g., asthma)
* Have a known metabolic disease (e.g., Type 1 diabetes)
* Are unable to exercise
* Are pregnant
* Less than 6 months post childbirth or stopped breastfeeding within the last month

Ages: 7 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population will be healthy children, adolescents and adults between the ages of 7-10 years, 12-16 years or 19-35 years of age. Participants will be recruited from the general population from online advertisements and media, targeting children, adolescents and adults residing in the Okanagan, British Columbia.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Cerebral blood flow | Experimental visit (1 day)
  Ultrasound assessment of the internal carotid artery blood flow

SECONDARY OUTCOMES:
Cerebral blood velocity | Experimental visit (1 day)
  Ultrasound assessment of the middle cerebral artery velocity
Beat-by-beat blood pressure | Experimental visit (1 day)
  Continuous assessment of mean arterial pressure responses
Saliva hormone concentrations | Experimental visit (1 day)
  Saliva specimen samples for the assessment of estrogen, progesterone, dehydroepiandrosterone and testosterone for the characterization of maturation status
Physical activity questionnaire | Experimental visit (1 day)
  Self report assessments of physical activity levels will be assessed
Anthropometrics: weight | Experimental visit (1 day)
  Body mass (kg) will be measured with electronic scales
Gas analysis | Experimental visit (1 day)
  The partial pressures of end-tidal carbon dioxide and oxygen will be sampled at the mouth from a fitted respiratory face mask.
Anthropometrics: height | Experimental visit (1 day)
  Stature standing and sitting height will be measured (cm).

CONTACTS AND LOCATIONS:
Overall Officials: Jared Baylis, MD, Principal Investigator — University of British Columbia

IPD SHARING:
Plan to Share IPD: Yes
Pseudonymized data from this study will be made available for sharing with other investigators, after publication of the study's key papers. Data will be shared through the Federated Research Data Repository (FRDR) (https://www.frdr-dfdr.ca/repo/). This is a secure data repository, which is searchable on the www, it is managed by Library Services. A digital object identifier (DOI) will be generated for datasets as they are deposited to the repository. Data will be stored in this repository for a minimum of 10 years or for 10 years from the last date of access.
Time Frame: Data will be stored in this repository for a minimum of 10 years or for 10 years from the last date of access.
Access Criteria: Data will be shared through the Federated Research Data Repository (FRDR) (https://www.frdr-dfdr.ca/repo/). This is a secure data repository, which is searchable on the www, it is managed by Library Services. A DOI will be generated for datasets as they are deposited to the repository.

REFERENCES:
- [Result] Ito S, Mardimae A, Han J, Duffin J, Wells G, Fedorko L, Minkovich L, Katznelson R, Meineri M, Arenovich T, Kessler C, Fisher JA. Non-invasive prospective targeting of arterial P(CO2) in subjects at rest. J Physiol. 2008 Aug 1;586(15):3675-82. doi: 10.1113/jphysiol.2008.154716. Epub 2008 Jun 19. PMID 18565992
- [Result] Fisher JA. The CO2 stimulus for cerebrovascular reactivity: Fixing inspired concentrations vs. targeting end-tidal partial pressures. J Cereb Blood Flow Metab. 2016 Jun;36(6):1004-11. doi: 10.1177/0271678X16639326. Epub 2016 Mar 21. PMID 27000209